CLINICAL TRIAL: NCT01704443
Title: Integrated Mindfulness for Provoked Vestibulodynia
Acronym: IMPROVED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H08-00885
Record Dates: First submitted 2012-08-24; First posted 2012-10-11 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Provoked Vestibulodynia
Keywords: provoked vestibulodynia; dyspareunia; vulvodynia; mindfulness; cognitive behavioural therapy
MeSH Terms: conditions — Dyspareunia; Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate treatment (Experimental): Women in the Immediate treatment arm will receive the Group Psychoeducational treatment in the next available group. There will be 8-9 womenper group and each session will be 2.25 hours in duration and there will be 4, bi-weekly sessions over the course of 2 months. Session content includes education about chronic pain, PVD, stress and sexual response, mindfulness practices, and cognitive techniques to notice thought patterns that contribute to increased pain.
  Interventions: Behavioral: Group Psychoeducational Treatment
- Waitlist Control- delayed treatment (Experimental): Women in the Waitlist Control arm will receive no treatment for a period of approximately 8 weeks. After the waitlist period they will receive the same Group Psychoeducational treatment as the participants in the immediate treatment arm of the study.
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: Group Psychoeducational Treatment — The Group Psychoeducational Treatment consists of treatment in small group format (8-9 women). Each session will be 2.25 hours in duration and there will be four, bi-weekly sessions over the course of 2 months. Session content includes education about chronic pain, PVD, stress and sexual response, mindfulness practices, and cognitive techniques to notice thought patterns that contribute to increased pain.
  Participants in the Waitlist Control Condition will receive this treatment at the end of the waitlist period (approximately 8 weeks)
  Arms: Immediate treatment
Other: Waitlist control — No treatment will be provided during the 8 week Waitlist control period
  Arms: Waitlist Control- delayed treatment

SUMMARY:
This study aims to test the efficacy of a 4-session intervention (Group psychoeducational treatment) using a randomized study design. Participants will be randomized in to 'immediate treatment' or 'waitlist control'. Women in the wait-list condition will receive the 4-session IMPROVED treatment, just as women randomized to the experimental group, after the end of their wait-list period.

ELIGIBILITY:
Inclusion Criteria:

* must be a patient at the British Columbia Centre for Sexual Medicine
* diagnosis of provoked vestibulodynia (PVD)
* 19 years of age or older
* premenopausal
* fluent in English

Exclusion Criteria:

* not at patient at the BC Centre for Sexual Medicine
* unprovoked vulvar pain, other pathology causing pain with penetration, or chronic pelvic pain
* being uncomfortable and unwilling to participate in a group setting.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity | one week pre-treatment to one week post treatment
  Pain intensity will be measured with the Q-tip test- a standard method of diagnosing vestibulodynia and assessing the pain associated with the diagnosis. The Q-tip test involves the physician lightly touching a Q-tip to specific areas around the vulvar vestibule while the patient indicates how much pain they feel on a scale from 0-10 in response to this provoked touch.
Long-term pain intensity | One week pre-treatment to 6 months post preatment
  Pain intensity will be measured with the Q-tip test- a standard method of diagnosing vestibulodynia and assessing the pain associated with the diagnosis. The Q-tip test involves the physician lightly touching a Q-tip to specific areas around the vulvar vestibule while the patient indicates how much pain they feel on a scale from 0-10 in response to this provoked touch

SECONDARY OUTCOMES:
Sexual Distress | One week pre-treatment, one week post treatment and 6-months follow up
  The investigators will examine women's self-reported sexual distress by administering the Female Sexual Distress Scale-Revised (Derogatis et al, 2008)

OTHER OUTCOMES:
Pain Catastrophising | one week pre-treatment, one week post treatment and 6-months follow-up
  The investigators will examine women's self-reported pain catastrophising by administering the Pain Catastrophizing Scale (Sullivan, Bishop & Pivik, 1995).
Pain hypervigilance | one week pre-treatment, one week post treatment and 6-months follow-up
  The investigators will examine women's self-report hypervigilance about pain by administering the Pain Vigilance and Awareness Questionnaire, McCracken, 1997)

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Centre for Sexual Medicine, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — http://www.obgyn.ubc.ca/SexualHealth/